CLINICAL TRIAL: NCT06791811
Title: A Comparative Study Between Opioids Free Anesthesia Using Dexmedetomidine and Lidocaine and Conventional Opioid Anesthesia on Stress Points Haemodynamics in Patients Undergoing Supratentorial Tumor Resection
Brief Title: A Comparative Study Between Opioids Free Anesthesia and Opioid Anesthesia in Patients With Supratentorial Tumor Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Sherif Alaa Embaby, Consultant of Anaesthesia, Surgical ICU and Pain management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MD-83-2024
Record Dates: First submitted 2024-09-07; First posted 2025-01-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Supra-tentorial Tumor
Keywords: Anaesthesia; dexmedetomidine; Craniotomy; Lidocaine; Opioid Free Anaesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid free Anaesthesia group (OFA) (Active Comparator): Prior to the induction of anesthesia the patients in OFA group will receive Dexmedetomidine and Lidocaine.
  Interventions: Other: OFA
- Opioid Anaesthesia group (OA). (Active Comparator): In the opioid anaesthesia group patients will receive fentanyl 2 μg/kg loading dose which will be prepared over 20 ml syringe and infused over 10 minutes prior to induction, Then after induction maintenance of analgesic infusion by fentanyl 0.5-1 μg/kg/h (200 micograms in 50 cc syringe with infusion rate 0.125-0.250ml/kg/h).Placebo (saline infusion) in 20 cc syringe with rate infusion rate 0.1 ml/kg/h.
  Interventions: Other: OA

INTERVENTIONS:
Other: OFA — Prior to the induction of anesthesia the patients in OFA group will receive Dexmedetomidine loading dose 1 μg/kg i.v. infusion, and Lidocaine loading dose 1.5 mg/kg i.v. infusion.
  The weight based doses of dexmedetomidine, lidocaine will be prepared in a 20 ml syringe and infused over 10 minutes prior to induction.
  Then after induction maintenance drugs will be infused as follow:
  Dexmedetomidine 0.25-0.5 μg/kg/h (200 micogram in 50cc syrige with infusion rate 0.125-0.250ml/kg/h), and Lidocaine 2mg/kg/h (400mg in 20cc syringe with infusion rate 0.1 ml/kg/h)
  Arms: Opioid free Anaesthesia group (OFA)
Other: OA — In the opioid anaesthesia group patients will receive fentanyl 2 μg/kg loading dose which will be prepared over 20 ml syringe and infused over 10 minutes prior to induction, Then after induction maintenance of analgesic infusion by fentanyl 0.5-1 μg/kg/h (200 micograms in 50 cc syringe with infusion rate 0.125-0.250ml/kg/h).Placebo (saline infusion) in 20 cc syringe with rate infusion rate 0.1 ml/kg/h.
  Arms: Opioid Anaesthesia group (OA).

SUMMARY:
Anesthesia for cranial surgeries is charactarized by periods of unpleasant stimuli interspersed with periods of low stimulation, which may compromise hemodynamic regulation.

Intraoperative and early postoperative episodes of hypertension during moments of strong stimulation can cause major consequences such as post craniotomy intracranial haemorrhage and vasogenic brain edema.

The use of powerful opioid analgesics like fentanyl and remifentanil in increasing doses for anaesthesia is a common practice among anesthesiologists.However, using strong opioids continuously or in bolus doses during surgery may result in postoperative hyperalgesia and higher analgesic need.

More recently, concerns have risen about impaired healing, immunosuppression , worsening of oncologic outcomes with systemic opioids and may affect conscious level at time of extubation (3).

Opioid-free anaesthesia(OFA) is increasingly gaining acceptance among anaesthesioligists. Its mainstay is based on a number of analgesic adjuvants that, when combined in small dosages, will produce effective anaesthesia with fewer side effects and a quicker recovery time than opioids. This approach, which combines several medications including dexmedetomidine, lidocaine, ketamine, ketorolac, and magnesium, has been used successfully in anaesthesia for bariatric procedures (3) . In cranial surgerie,OFA has been mainly used in pilot studies and case reports and their main focus was postoperative opioid consumption and not intraoperative haemodynamics.(4).

Dexmedetomidine which is a highly selective 2-adrenoceptor agonist has positive effects as anesthetic adjuvant.It has sedative, anxiolytic, and analgesic effects with little impact on respiratory drive, Dexmedetomidine analgesic properties are less potent than opioids, despite the fact that preoperative intravenous dexmedetomidine administration is linked to a reduction in postoperative pain intensity, analgesic intake, and nausea.

According to reports, intravenous lidocaine possesses analgesic, anti-hyperalgesic, and anti-inflammatory actions by inhibition of the priming of resting neutrophilic granulocytes which may reduce the liberation of superoxide anions a common pathway of inflammation. It has potentials for brain protections as it reduces cerebral oxygen consumption, cerebral blood volume and flow .Moreover ,it decreases the intracranial pressure and consequently results in brain relaxation.

The addition of a scalp block to general anaesthetic during craniotomies might lessen the discomfort associated with scalp incision and pin application, as well as the need for analgesics such as opioids or anaesthesia adjuvants, encouraging early recovery for neurological evaluation. The usage of this block has increased as a result of recent developments in neurosurgery, particularly awake craniotomy.

To our knowledge ,the effects of continuous intravenous lidocaine and dexmedetomidine infusion on hemodynamics, brain relaxation and surgeon satisfaction in adult patients undergoing cranial surgeries for tumor excision without the use of opioids, however, have not been studied.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ι and II.
2. Patients undergoing resection of supratentorial tumors in supine position.
3. Age (18-50) years.
4. Both sexes.

Exclusion Criteria:

1. Impaired renal functions.
2. Uncontrolled systemic hypertension(patients with sustained elevated blood pressure more than 140/90).
3. Cardiac arrhythmias (any rhythm other than normal sinus rhythm and sinus tachycardia).
4. Heart failure(impaired cardiac contractility ,EF less than 45%.).
5. Patients receiving more than 2 units of blood during surgery.
6. Patients with large masses and expected severe increase in ICP.
7. Patients requiring vasopressors infusion.
8. The need for postoperative ventilation at the end of study.
9. Glasgow coma scale less than 14.
10. History of allergy to the study drugs.
11. Surgeries lasting more than 4 hours.
12. Pregnancy.
13. Bronchial asthma.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patents experiencing a change in mean arterial pressure at time of Burr Hole | During the bur hole procedure around 20-30 minutes
  Percentage of patients experiencing a change in mean arterial pressure at time of Burr Hole ( Time Frame :During Burr hole surgery) Defined as recording an increase of the mean arterial blood pressure by more than 20% from baseline readings at time of burr hole.

CONTACTS AND LOCATIONS:
Overall Officials: Rania Samir, professor, Study Director — Department of anaesthesia
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All the data related to the study would be available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 month after the study is published.
Access Criteria: Any relatable study with an official request.

REFERENCES:
- [Background] Chandra S, Pryambodho P, Omega A. Evaluation of continuous intravenous lidocaine on brain relaxation, intraoperative opioid consumption, and surgeon's satisfaction in adult patients undergoing craniotomy tumor surgery: A randomized controlled trial. Medicine (Baltimore). 2022 Sep 9;101(36):e30216. doi: 10.1097/MD.0000000000030227. PMID 36086723
- [Background] Syeda S, Palaniswamy SR, Sriganesh K. Opioid Free Analgesia With Dexmedetomidine for Craniotomy in an Obese Patient With Obstructive Sleep Apnea and Difficult Airway. Asian J Anesthesiol. 2020 Jun 1;58(2):76-77. doi: 10.6859/aja.202006_58(2).0007. Epub 2020 Jul 24. No abstract available. PMID 33171574